CLINICAL TRIAL: NCT05451420
Title: The Efficacy and Safety of Inactive Hepatitis B Surface Antigen (HBsAg) Carriers (IHCs) Treated With Pegylated Interferon α2b Based Intervention Therapy(HBsAg Positive, HBeAg Negative, ALT Normal, HBsAg ≤ 1500IU/ml, HBV DNA ≤ 2000IU/ml)
Brief Title: Inactive HBsAg Carriers (IHCs) Treated With Pegylated Interferon α2b Based Intervention Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Henan Provincial People's Hospital (Other)
Collaborators: Xiamen Amoytop Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HenanPPHGRK
Record Dates: First submitted 2022-06-23; First posted 2022-07-11 (Actual); Last update posted 2022-07-13 (Actual); Status verified 2022-06

CONDITIONS: Chronic Hepatitis B
Keywords: inactive hepatitis B virus carriers; HBsAg clearance; peginterferon alpha 2b; Intervention treatment
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — Long-Term Synaptic Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): PegIFN α- 2b monotherapy, 180 μg/ week, 68 weeks of treatment, 24 weeks of follow-up after drug withdrawal
  Interventions: Drug: PegIFN α- 2b
- Group B (Active Comparator): Patients had a lead-in period of 16 weeks before baseline, pegifn α- 2b single drug treatment for 24 weeks, 4 weeks after drug withdrawal, 16 weeks of introduction period, pegifn α- 2b was followed up for 24 weeks. The plan of the induction period is as follows: 1) from the first day of the induction period, GM-CSF is injected subcutaneously ® one hundred μg/ piece, produced by Xiamen Tebao Bioengineering Co., Ltd.), 100 μg/ day, 5 consecutive days, one cycle every 4 weeks, 4 consecutive cycles. 2) On the third day of the induction period, recombinant hepatitis B vaccine (Saccharomyces cerevisiae) (1.0ml/HBsAg 60 per dose) was injected subcutaneously μg. Shenzhen Kangtai Biological Products Co., Ltd.), 60 μ g. Once every 4 weeks for 4 consecutive cycles, the course of treatment was 68 weeks, and the patients were followed up for 24 weeks.
  Interventions: Drug: PegIFN α- 2b

INTERVENTIONS:
Drug: PegIFN α- 2b — Adjuvant immunotherapy with GM-CSF and Hepatitis B vaccine
  ；GM-CSF（100 μg/ piece, produced by Xiamen Tebao Bioengineering Co., Ltd）；Hepatitis B vaccine（Each 1.0ml/HBsAg60 μ g. Shenzhen Kangtai Biological Products Co., Ltd）
  Other Names: pegbin ® 180μg，produced by Xiamen Tebao Bioengineering Co., Ltd.

SUMMARY:
A single center, randomized controlled trial design was used to select patients with chronic hepatitis B in the immune control period (HBsAg positive, HBeAg negative, normal ALT, HBsAg ≤ 1500iu/ml, HBV DNA ≤ 2000iu/ml) to enter the study, and to compare the feasibility, effectiveness and safety of pegylate combined with Granulocyte-macrophage colony stimulating factor, high-dose hepatitis B vaccine and pegylate monotherapy in the treatment of patients with chronic hepatitis B in the immune control period

DETAILED DESCRIPTION:
Explore the efficacy, safety and related influencing factors of intervention therapy based on PegIFN α- 2b in inactive hepatis B surface antigen (HBsAg) carriers (IHCs), and compare pegifn α- 2b combined with granulocyte macrophage stimulating factor (GM-CSF), high-dose hepatitis B vaccine and pegifn α- 2B feasibility, efficacy and safety of monotherapy for IHCs.The IHCs patients were randomly divided into two groups (group A: pegifn α- 2b single drug group, group B: pegifn α- 2b combined with GM-CSF and high-dose hepatitis B vaccine group). To start applying pegifn α- 2B was the baseline, treatment for 68 weeks, followed up for 24 weeks after drug withdrawal. Patients in group B used GM-CSF and vaccine introduction for 16 weeks before baseline.The HBsAg clearance rate and related influencing factors of the two groups at 68 weeks were analyzed.

ELIGIBILITY:
Inclusion Criteria:

* age 18 to 65 years;
* HBsAg seropositive status for more than 6 months prior to enrollment;
* never received treatment with any form of nucleos(t)ide analogues (NAs) or interferon before enrollment;
* Serum HBsAg ≤1500 IU/mL;
* HBeAg negative with or without HBeAb positive;
* Serum HBV DNA ≤2000IU/ml IU/mL;
* normal ALT levels;
* normal white blood cell and platelet counts;
* abdominal computed tomography or B-ultrasound showed no cirrhosis, splenomegaly or ascites.

Exclusion Criteria:

* Participants with other hepatotropic viruses or human immunodeficiency virus co-infection
* other chronic non-viral liver diseases or decompensated liver diseases
* tumours
* drug abuse
* severe psychiatric disease
* uncontrolled thyroid disease or diabetes
* pregnancy or lactation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
HBsAg clearance at the end of 68 weeks of treatment | 68 weeks of treatment
  To determine the response rate will be evaluated by HBsAg loss defined as HBsAg level lower than 0.05 IU/ml after 48 week treatment, compared with control group.

SECONDARY OUTCOMES:
HBsAg level and the decreasing extent of HBsAg level | baseline，12 weeks, 24 weeks, 44 weeks，56 weeks， 68weeks，80 weeks，92weeks of treatment
  To assessment the decreasing level and difference of HBsAg levels in different treatment groups
HBsAg seroconversion rate | 68 weeks of treatment
  To assessment the HBsAg seroconversion rate in different treatment groups

OTHER OUTCOMES:
HBsAg clearance and seroconversion rate of PEG IFN based immunoadjuvant combined therapy | baseline，12 weeks, 24 weeks, 44 weeks，56 weeks， 68weeks，80 weeks，92weeks of treatment
  To assessment the HBsAg clearance and seroconversion rate of immunoadjuvant combined therapy on 68 weeks' curative effect

CONTACTS AND LOCATIONS:
Overall Officials: Jia Shang, Study Chair — Henan Provincial People's Hospital
Locations (1):
- Henan Provincial People's Hospital, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: Yes
After publication
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: End of study
Access Criteria: Editors and reviewers of contributing magazines

REFERENCES:
- [Derived] Ning H, Li K, Peng Z, Jin H, Zhao H, Shang J. The efficacy and safety of pegylated interferon alpha-2b-based immunotherapy for inactive hepatitis B surface antigen carriers. Eur J Gastroenterol Hepatol. 2023 Oct 1;35(10):1216-1223. doi: 10.1097/MEG.0000000000002627. Epub 2023 Aug 14. PMID 37577817